CLINICAL TRIAL: NCT04118673
Title: Secondary Care - Prescribing Lifestyle Adjustments for Cardiovascular Health (Phase II)
Brief Title: Secondary Care - Prescribing Lifestyle Adjustments for Cardiovascular Health (S-PLAC 2)
Acronym: S-PLAC 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: CV-19 pandemic
Sponsor: University of South Wales (Other)
Collaborators: Public Health Wales (Other Government); Cwm Taf University Health Board (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 260481
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Health Behavior
MeSH Terms: conditions — Cardiovascular Diseases; Health Behavior

STUDY DESIGN:
Intervention Model Description: The study is an interventional controlled observational study based in the Secondary care setting. Control groups will be utilized through the mechanism of wait-listing the enrolment of recruitment centres into the study.
  Mixed methods will be used for both data collection and analysis. Historical clinical participant data (pre-intervention) will be collected by the PI. data will be collected immediately after the consultation and at 3 months post intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Standard Care) (No Intervention): Standard care during consultations. Advice and guidance offered by clinicians verbally and sometimes the addition of leaflets or a referral.
- Intervention (Standard Care plus Lifestyle prescription - LRx) (Experimental): Standard care during consultations with the addition of a physical lifestyle prescription. Advice and guidance will be offered by clinicians verbally, whilst being supported with a lifestyle prescription and a possible referral if required.
  Interventions: Behavioral: Lifestyle Prescription (LRx)

INTERVENTIONS:
Behavioral: Lifestyle Prescription (LRx) — Standard care during consultations with the addition of a physical lifestyle prescription
  Arms: Intervention (Standard Care plus Lifestyle prescription - LRx)

SUMMARY:
Prescribing lifestyle changes to patients who have cardiovascular disease (CVD) may be an extremely cost effective mechanism of improving health individually and for the NHS. Positive lifestyle changes such as improved diet, increased physical activity, quitting smoking and reducing alcohol consumption have been proven to reform the health status of individuals with CVD. S-PLAC 2 is a phase II study to determine the efficacy of a lifestyle prescription (L℞) in patients and healthcare practitioners in a secondary care setting (i.e. hospital clinics/wards).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Able and willing to provide written informed consent
* Understands written and spoken English
* Either an in/out- patient of Cardiology

Exclusion Criteria:

* Participant is unwilling or unable to provide written informed consent
* Participant is pregnant
* Participant has a drug dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
A prescription (LRx) being issued during a consultation | During month 7 of the study
  Number of so-signed prescription (LRx) forms. Total number of forms to be co-signed = 60
Patient view of the prescription (LRx) and consultation Questionnaire | During month 7 of the study
  Completed study questionnaires. Total number of questionnaires to be completed = 120. Responses will be recorded to gain feedback from the patient participants regarding their thoughts and feelings of their consultation with and without the intervention of the prescription (LRx).
  Scale: 7 (minimum) to 41 (maximum). A lower value represents a better (more positive) outcome.
Healthcare practitioner (HCP) view of the prescription (LRx) and consultation questionnaire. | During month 7 of the study
  Completed clinician questionnaire. Total number of questionnaires to be completed = 6. Responses will be recorded to gain feedback from the clinicians regarding their thoughts and feelings of their consultations with and without the intervention of the prescription (LRx).
  Sections:
  Section 1 scale: 9 to 54 (a lower score represents a better, more positive outcome) Section 2 scale: 8 to 48 (a lower score represents a better, more positive outcome) Section 3 scale: 6 to 36 (a lower score represents a better, more positive outcome) Total score available: 23 to 138

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Wales, Pontypridd, United Kingdom

IPD SHARING:
Plan to Share IPD: No